CLINICAL TRIAL: NCT02262390
Title: Comparison of Different Partner Notification Strategies After Antenatal Syphilis Screening
Brief Title: Syphilis Treatment of Partners Trial
Acronym: STOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other)
Responsible Party: Principal Investigator, Infectious Diseases Institute, Head of Prevention Care & Treatment, IDI, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ST/0109/14
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Syphilis Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (Active Comparator): Partner notification slip is given to the pregnant female participant on the day she receives her syphilis test results to give to their sexual partner encouraging them to come to the STI clinic and be screened for syphilis. The partner notification slip will have a code number, but no identifiable features (no names).
  Interventions: Procedure: Partner Notification Reminders
- SMS reminders and notification slip for partner screening (Active Comparator): Participants will receive weekly SMS reminders to encourage their partners to attend the STI clinic for syphilis testing for up to 8 weeks after initial positive syphilis test for the participant. The participant ID number will be written on both the notification paper which partners should bring in with them and on the SMS reminders.
  Interventions: Procedure: Partner Notification Reminders
- Phone call reminders and notification slip for partner scree (Active Comparator): Participants will receive weekly phone call reminders to encourage their partners to attend the STI clinic for syphilis testing for up to 8 weeks after initial positive syphilis test for the participant. The participant ID number will be written on both the notification paper which partners should bring in with them and be given to the participant when the nurse calls.
  Interventions: Procedure: Partner Notification Reminders

INTERVENTIONS:
Procedure: Partner Notification Reminders — For all 3 arms, the following will be done:
  * All participants will have an antenatal clinic visit every 4 weeks until delivery.
  * All notification slips will be duplicate; one given to the mother and one held in the clinic. The study ID number will be documented on the slip. On partner return the slips will be matched and used to link mothers with male returning partners.
  * Partner participant test result will be linked to the patient using the participant ID number in the lab. Partners will be tested using a rapid treponemal antibody test.

SUMMARY:
2.1 Primary Study Hypothesis In sub-Saharan Africa, between 2.5-17% of pregnant women are infected with syphilis [1]. It is estimated that 53-82% of women with untreated syphilis had adverse outcomes compared to only 10-21% of uninfected women[2]. The investigators and others have shown that syphilis screening integrated into an HIV antenatal clinic with prevention of mother to child transmission (PMTCT) is highly accepted with excellent uptake. Unfortunately, the minority of male partners come in for testing and treatment (1%-27%) which has important implications for the roll-out of rapid syphilis testing and the inability to detect reinfection with treponemal antibody test as the test will remain positive despite treatment. The investigators hypothesize that sending an SMS reminder or a telephone call reminder by a health care worker will be more effective than a standard notification slip given to women to bring male partners to antennal clinic for testing and treatment.

DETAILED DESCRIPTION:
Title: Comparison of Different Partner Notification Strategies after Antenatal Syphilis Screening Short Title: Syphilis Treatment of Partners (STOP) Trial Objectives: Primary For pregnant women who test rapid syphilis test positive; to compare the proportion of male partners who report to the clinic for syphilis testing (and treatment) when the women are given only partner notification slips (standard of care) compared to a notification slip plus a weekly automated SMS reminder OR a notification slip plus a weekly nurse phone call reminder.

Secondary

* To compare the proportion of male partners who test positive for syphilis when they report to the clinic after receiving notification in the three groups via their pregnant partners.
* To compare the proportion of male partners who undergo treatment among the three groups.
* To explore factors associated with reporting/not reporting after notification.
* To compare birth outcomes (congenital syphilis, stillbirths, neonatal deaths, preterm or low birth weight) between the three arms (self-reported by women).
* To assess time from syphilis point of care (POC) test to treatment in mothers who test syphilis positive using a rapid treponemal antibody kit.
* To compare the proportion of women who have a 4-fold decrease in RPR titer by intervention arm in each arm at post natal visit.

Study Population and sample size: • Pregnant women from 14years and above reporting to antenatal and subsequently postnatal clinics at the Infectious Disease Institute, Mulago Hospital (antenatal and STI clinics), and Kasangati Health Center IV in Kampala, Uganda who screen positive by rapid treponemal antibody test.

* Male sexual partners to these enrolled syphilis positive pregnant mothers.
* 876participants will be enrolled. Study Design: Individual patient randomized open-label clinical trial of syphilis partner notification interventions.

Study Duration: Approximately 24 months

Endpoints:

Primary:

1) Proportion of male partners who present at clinic and receive syphilis testing

Secondary:

1. Male partners tested (standard vs. intervention in 3 arm randomization)
2. Proportion of male partners who test positive for syphilis when they report to the clinic after notification.
3. Proportion of syphilis positive male (tested by syphilis POCT) partners who undergo treatment among the three groups.
4. Factors associated with partners reporting/not reporting after notification.
5. Syphilis infected pregnant women re-tested in 3rd trimester with a 4-fold dilutional titer decrease in RPR (by standard vs. intervention arm)
6. Mother reported birth outcomes (by standard vs. intervention arm) Subject Participants: Pregnant women testing positive for syphilis at the antenatal clinics and their partners.

Description of Study Design: This is a prospective clinical trial in which pregnant syphilis positive women (tested by rapid treponemal antibody kit) will be randomized to one of three arms to notify participants to bring their sexual partners at risk for syphilis for syphilis screening and treatment. Women will be randomized in a 1:1:1 ratio to one of the following three strategies: A) To receive a notification slip per the Ministry of Health standard B) to receive a notification slip plus an SMS reminder or C) to receive a notification slip plus standardized nurse/clinician initiated phone call.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the following inclusion criteria in order to be eligible to participate:

* Pregnant women
* Treponemal antibody rapid positive test
* Age> 14 years
* Written informed consent
* Known sexual partner
* Access to cell phone and willing and able to use and receive SMS or phone calls In the Uganda guidelines (section 9.3 Mature and Emancipated Minors), "mature minors are individuals 14-17 years of age who have drug or alcohol dependency or a sexually transmitted infection; Mature minors may independently provide informed consent to participate in research if in the view of the IRC the research is not objectionable to parents or guardian (established by the IRC with evidence from the community); and b) The research protocol include clear justification for targeting mature and emancipated." This protocol will recruit pregnant women with a sexually transmitted infection in an intervention with minimal risk and with the potential to prevent future reinfection.

Exclusion Criteria:

* Any subjects meeting any of the following exclusion criteria at baseline will be excluded from study participation:

  * Illiterate and unable to read a text message
  * Inability to use a mobile phone
  * Patients with confirmed neuro syphilis treated with IV Benzyl penicillin

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1752 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of male partners who present at clinic and receive syphilis testing | 2 years
  Proportion of male partners who present at clinic and receive syphilis testing

SECONDARY OUTCOMES:
Male partners tested (standard vs. intervention in 3 arm randomization) | 2 years
  Male partners tested (standard vs. intervention in 3 arm randomization)
Proportion of male partners who test positive for syphilis when they report to the clinic after notification. | 2 years
  Proportion of male partners who test positive for syphilis when they report to the clinic after notification.
Proportion of syphilis positive male (tested by syphilis POCT) partners who undergo treatment among the three groups. | 2 years
  Proportion of syphilis positive male (tested by syphilis POCT) partners who undergo treatment among the three groups.
Factors associated with partners reporting/not reporting after notification. | 2 years
  Factors associated with partners reporting/not reporting after notification.
Syphilis infected pregnant women re-tested in 3rd trimester with a 4-fold dilutional titer decrease in RPR (by standard vs. intervention arm) | 2 years
  Syphilis infected pregnant women re-tested in 3rd trimester with a 4-fold dilutional titer decrease in RPR (by standard vs. intervention arm)
Mother reported birth outcomes (by standard vs. intervention arm) | 2 years
  Mother reported birth outcomes (by standard vs. intervention arm)

CONTACTS AND LOCATIONS:
Overall Officials: Yuka C Manabe, MD, Study Chair — Johns Hopkins University
Locations (1):
- Infectious Diseases Institute, Kampala, Kampala, Uganda

REFERENCES:
- [Derived] Nakku-Joloba E, Kiguli J, Kayemba CN, Twimukye A, Mbazira JK, Parkes-Ratanshi R, Birungi M, Kyenkya J, Byamugisha J, Gaydos C, Manabe YC. Perspectives on male partner notification and treatment for syphilis among antenatal women and their partners in Kampala and Wakiso districts, Uganda. BMC Infect Dis. 2019 Feb 6;19(1):124. doi: 10.1186/s12879-019-3695-y. PMID 30727950